CLINICAL TRIAL: NCT06290089
Title: Pre-Study of Wild Type Enterotoxigenic E. Coli (ETEC) Strain for Verification of a Planned Challenge Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scandinavian Biopharma AB (Industry)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OEV-131
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: ETEC Diarrhea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETEC strain (Other): Each enrolled subject will receive a single administration of the challenge dose
  Interventions: Other: Enterotoxigenic E. coli (ETEC) strain

INTERVENTIONS:
Other: Enterotoxigenic E. coli (ETEC) strain — Challenge strain

SUMMARY:
This was an open-label, single-site pre-study designed to evaluate the safety, tolerability, and infectivity of wild-type Enterotoxigenic Escherichia coli (ETEC) strain E24377A in healthy adults. The aim was to estimate the incidence of moderate and severe diarrhea following oral challenge with approximately 4 × 10⁹ colony forming units (cfu) of the strain.

A total of 23 participants were enrolled and monitored in an inpatient setting after receiving a single challenge dose. Clinical signs, symptoms, and stool output were assessed over 120 hours. This challenge model was developed to support a future controlled human infection study (CHIM) evaluating an oral inactivated ETEC vaccine.

DETAILED DESCRIPTION:
This was an open-label, single-center pre-study designed to evaluate the safety, tolerability, and infectivity of wild-type Enterotoxigenic Escherichia coli (ETEC) strain E24377A in healthy adults. The goal was to estimate the incidence of moderate and severe diarrhea following challenge with approximately 4 × 10⁹ colony forming units (cfu) of the strain. This challenge model was intended to inform a subsequent controlled human infection model (CHIM) study assessing the efficacy of the oral inactivated tetravalent ETEC vaccine ETVAX® (containing LCTBA and dmLT).

Up to 30 healthy adult subjects were planned to be enrolled; 23 were ultimately challenged at the Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health in Baltimore, Maryland, USA. Participants underwent screening, then entered an inpatient unit on Day -1. On Day 1, they received a single oral dose of strain E24377A (lot 0807) suspended in 30 mL sodium bicarbonate buffer, preceded by 120 mL of buffer to reduce gastric acidity.

During the inpatient period, subjects were monitored at least three times daily for vital signs, signs and symptoms of ETEC illness, and stool output. All stools were collected, weighed, graded, and cultured. Stools were graded on a 5-point scale: Grade 1 = firm/formed; Grade 2 = soft/formed; Grade 3 = thick liquid; Grade 4 = thin liquid; Grade 5 = clear/watery. Loose stools were defined as Grade 3-5.

Diarrhea was defined as ≥2 loose stools (Grade 3-5) within a 24-hour period. Severity was categorized as:

Mild: 2-3 Grade 3-5 stools and ≤400 g in 24 h

Moderate: 4-5 Grade 3-5 stools or >400-800 g

Severe: ≥6 Grade 3-5 stools or >800 g

An independent adjudication committee determined whether episodes were attributable to ETEC and whether participants met the primary endpoint. Participants received ciprofloxacin 500 mg twice daily for 3 days starting on Day 6, or earlier if needed. Discharge occurred after meeting microbiological and clinical criteria, with follow-up visits on Day 29 (clinic) and Day 180 (phone).

Secondary and exploratory endpoints included stool frequency and weight, symptom scores, microbiological shedding, and immunologic assessments (serum, fecal, and ALS IgA/IgG, memory B cells, transcriptomics, and biomarkers of intestinal/systemic inflammation). Safety endpoints included adverse events through Day 29 and serious adverse events through Day 180.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between 18 and 50 years of age, inclusive, at the time of signing the informed consent.
2. General good health, without clinically significant medical history, physical examination findings or clinical laboratory abnormalities per clinical judgment of PI.
3. Negative pregnancy test at screening and prior to challenge for people of childbearing potential. People of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. People of childbearing potential unable to bear children must have this documented (e.g. tubal ligation or hysterectomy) or must have negative pregnancy tests at screening and prior to challenge.
4. Willingness to participate in the study after all aspects of the protocol have been explained and written informed consent obtained.
5. Completion of a training session and demonstrated comprehension of the protocol procedures and knowledge of ETEC associated illness by passing a written examination (70% pass score).
6. Availability for the study duration, including planned follow-up visit/contact.

Exclusion Criteria:

1. Presence of a significant medical or psychiatric condition which in the opinion of the investigator precludes participation in the study, including gastrointestinal disease (gastritis, irritable bowel disease as suggested by Rome III criteria or medical diagnosis, inflammatory bowel disease). Some medical conditions which are adequately treated and stable would not preclude entry into the study. These conditions might include stable asthma controlled with inhalers or mild hypertension stably controlled.
2. Significant abnormalities in screening haematology, or serum chemistry as determined by PI.
3. Presence in the serum of HIV antibody, HBsAg, or HCV antibody with confirmation of infection (e.g. by HCV PCR).
4. Evidence of IgA deficiency (serum IgA < 7 mg/dl or limit of detection of assay).
5. Evidence of current alcohol or drug dependence.
6. Subjects whose Body Mass Index (BMI) is less than 19.0 or greater than 37.0 (kg/m2).
7. Recent vaccination or receipt of an investigational product (within 30 days before challenge) or intended vaccination or receipt of investigational products until 60 days after challenge, with the exception of licensed vaccine for influenza or SARS-CoV-2 vaccination that may be given up to 7 days prior to challenge.
8. Positive test for SARS-CoV-2 at arrival to the unit on the day of in-patient admission.
9. Intention to donate blood or blood products within one month following the completion of study participation (note: The Red Cross will not allow blood donations for 1 year following participation in an investigational research study).
10. Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the safety of the study, or the results of the study.
11. Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
12. Regular (≥ weekly) use of laxatives, antacids, or other agents to lower stomach acidity.
13. Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the challenge or planned use during the active study period. Use of inhaled or topical steroids may be permitted per PI discretion.
14. History of microbiologically confirmed ETEC infection in the last 3 years.
15. Occupational handling of ETEC currently, or in the past 3 years.
16. Travel to countries where ETEC infection is endemic (most of the developing world) within two years prior to dosing OR visit for > two months in ETEC endemic countries during the last 10 years, OR planned travel to endemic countries prior to study day 180.
17. Vaccination for or ingestion of ETEC, cholera, or LT toxin within 5 years prior to dosing.
18. Use of antibiotics during the 14 days before challenge dosing or proton pump inhibitors, H2 blockers or antacids within 48 hours prior to challenge dosing.
19. History of diarrhea in the 7 days prior to challenge (outpatient diarrhea is defined as ≥ 3 unformed (grade 3 or greater) loose stools in 24 hours).
20. Known allergy to two of the three following antibiotics: ciprofloxacin, amoxicillin, and/or azithromycin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ETEC Strain
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all subjects who have been challenged with E24377A (regardless if the whole intended challenge dose was ingested or a subject vomited just after ingestion) and have available data. The Full Analysis Set will be included in analyses of all endpoints.
Groups:
- Challenge Dose Only Group: A total of 23 subjects were enrolled in this arm. All participants received a single oral challenge dose of ETEC strain E24377A . The objectives are to evaluate the moderate and severe diarrhea attack rate, the safety and the immunogenicity. No prior vaccination was administered in this group.
Arm/Group | Challenge Dose Only Group
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: year] — Description of scale
  year | 39 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 7
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 23
Height [Mean (Standard Deviation); unit: cm] | 175.70 (10.53)
Weight [Mean (Standard Deviation); unit: kg] | 86.56 (15.46)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate and Severe Diarrhea
Description: Defined as ≥ 4 grade 3-5 stools or > 400 grams of grade 3-5 stools passed within a rolling 24-hour period, deemed attributable to ETEC
Time Frame: 120 hours post-challenge
Population: The Full Analysis Set includes all subjects who were challenged with E24377A (regardless of whether the whole intended challenge dose was ingested, or a subject vomited just after ingestion) and had available data. The Full Analysis Set was to be included in analyses of all endpoints
Measure: Number; unit: participants moderate or severe diarrea
Arm/Group | ETEC Strain
Number analyzed (Participants) | 23
participants moderate or severe diarrea | 17

2. Primary Outcome: Subjects Developing Moderate-to-Severe Diarrhea Following Oral Challenge
Description: Each stool was to be graded according to the following scale:
  Grade 1 = firm, formed Grade 2 = soft but still formed Grade 3 = thick liquid Grade 4 = thin liquid Grade 5 = clear or translucent, watery A loose stool was defined as a Grade 3-5 stool. Diarrhea was defined as passing at least 2 loose (Grade 3-5) stools within a 24-hour period.
  Diarrhea severity was to be assigned according to the scale in Table 4.
  Diarrhea Rating Scale:
  Mild 2-3 Grade 3-5 stools in 24 hours and ≤ 400 grams of Grade 3-5 stools passed in a 24- hour period Moderate 4-5 Grade 3-5 stools in 24 hours or > 400-800 grams of Grade 3-5 stools passed in a 24-hour period Severe ≥ 6 Grade 3-5 stools in 24 hours or > 800 grams of Grade 3-5 stools passed in a 24-hours period.
Time Frame: up to 120 hours post-challenge
Population: The Full Analysis Set includes all subjects who were challenged with E24377A (regardless of whether the whole intended challenge dose was ingested, or a subject vomited just after ingestion) and had available data.
Measure: Number (95% Confidence Interval); unit: percentage of subject with MSD
Arm/Group | Challenge Dose Only Group
Number analyzed (Participants) | 23
percentage of subject with MSD | 74 [51.6 to 89.8]

ADVERSE EVENTS:
Time Frame: Unsolicited AEs were collected until Day 29, and SAEs and adverse events of special interest (AESIs) were collected until Day 180. Approximately 6 months after challenge, allsubjects will have a follow-up contact by telephone to inquire about the occurrence of any new chronic illnesses or serious adverse events
Description: * Adverse events, includes all adverse events observed after challenge, regardless of their relationship to the challenge strain
  * Serious adverse events (SAEs) occurring during the 6 months of the study (from the time of challenge)
Arm/Group | ETEC Strain
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 14/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETEC Strain (N=23)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 3 (4)
Eructation (Gastrointestinal disorders) | 3 (4)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dyspesia (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vormiting (Gastrointestinal disorders) | 1 (1)
Blood presure increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Muscel spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Presyncope (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The target enrollment was 30 participants, the data from the 23 enrolled subjects provided sufficient insight into the expected attack rates across diarrhea severity levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT06290089/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT06290089/SAP_001.pdf